CLINICAL TRIAL: NCT06996834
Title: A Randomized Controlled Trial of High-Velocity Nasal Insufflation (HVNI) Versus Noninvasive Ventilation (NIV) for Acute Respiratory Failure of Community-Acquired Pneumonia (CAP).
Brief Title: Noninvasive Support Methods for Acute Respiratory Failure of Community-acquired Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Shaddad, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 307052025
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Community-acquired Pneumonia; Community-Acquired Infections
Keywords: CAP; NIV; HVNI
MeSH Terms: conditions — Community-Acquired Pneumonia; Community-Acquired Infections | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, controlled, parallel-group clinical trial. Participants will be randomly assigned in a 1:1 ratio to receive either high-velocity nasal insufflation (HVNI) or noninvasive ventilation (NIV). Each participant will remain in their assigned intervention group for the duration of the study. The primary objective is to compare the efficacy of HVNI versus NIV in managing acute exacerbations of community-acquired pneumonia (CAP) by assessing treatment failure rates within 48 hours, defined as the need for intubation or death. Secondary outcomes include changes in gas exchange parameters, patient comfort levels, ICU length of stay, and 28-day mortality rates.
Who Masked: Outcomes Assessor
Masking Description: This is an open-label trial wherein participants, care providers, and investigators are aware of the assigned interventions. To minimize assessment bias, outcome assessors responsible for evaluating primary and secondary endpoints will remain blinded to treatment allocations throughout the study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Invasive Ventilation (NIV) (Experimental): Intervention:
  Participants in this arm will receive non-invasive ventilation using bilevel positive airway pressure (BiPAP) delivered via a full-face mask to support ventilation in patients with acute hypoxemic respiratory failure due to community-acquired pneumonia (CAP).
  Interventions: Device: Non-Invasive ventilation (NIV)
- High velocity nasal insufflation (HVNI) (Experimental): Intervention:
  Participants in this arm will receive high-velocity nasal insufflation therapy, a type of high-flow nasal cannula (HFNC) therapy that delivers heated and humidified oxygen at high flow rates to support patients with acute hypoxemic respiratory failure resulting from community-acquired pneumonia (CAP).
  Interventions: Device: High Velocity Nasal Insufflation

INTERVENTIONS:
Device: Non-Invasive ventilation (NIV) — Participants in this arm will receive noninvasive ventilation using bilevel positive airway pressure (BiPAP) delivered via a full-face mask to support ventilation in patients with acute hypoxemic respiratory failure due to CAP.
  Other Names: BI-level Positive airway pressure ventilation (BIPAP)
  Arms: Non-Invasive Ventilation (NIV)
Device: High Velocity Nasal Insufflation — Participants in this arm will receive high-velocity nasal insufflation therapy, a type of high-flow nasal cannula (HFNC) therapy that delivers heated and humidified oxygen at high flow rates to support patients with acute hypoxemic respiratory failure resulting from community-acquired pneumonia (CAP).
  Other Names: High velocity nasal cannula; Vapotherm delivery system
  Arms: High velocity nasal insufflation (HVNI)

SUMMARY:
This randomized controlled trial aims to compare the efficacy and safety of high-velocity nasal insufflation (HVNI) versus standard noninvasive ventilation (NIV) in adult patients experiencing acute exacerbations of community-acquired pneumonia (CAP) accompanied by hypoxemic respiratory failure. The primary focus is on assessing treatment failure within 48 hours, defined as the need for intubation or death. Secondary outcomes include evaluations of gas exchange parameters, patient comfort levels, duration of ICU stay, and 28-day mortality rates.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a significant contributor to acute hypoxemic respiratory failure, often necessitating ventilatory support. Noninvasive ventilation (NIV) has been a conventional approach; however, it can be associated with patient discomfort and varying success rates. High-velocity nasal insufflation (HVNI) presents an alternative, delivering heated and humidified oxygen at high flow rates, which may improve oxygenation and patient tolerance.

This study is designed as a prospective, randomized, open-label, parallel-group trial involving 100 adult patients diagnosed with CAP-induced hypoxemic respiratory failure. Participants will be randomly assigned to receive either high-volume non-invasive ventilation (HVNI) or non-invasive ventilation (NIV). The primary endpoint is treatment failure within 48 hours post-randomization, characterized by the necessity for endotracheal intubation or mortality. Secondary endpoints encompass changes in arterial blood gas measurements, patient-reported comfort scores, length of ICU stay, and 28-day mortality rates.

By systematically comparing HVNI and NIV in this patient population, the study seeks to determine whether HVNI offers a viable and potentially superior alternative to traditional NIV methods in managing acute respiratory failure due to CAP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical and radiographic diagnosis of CAP
* Respiratory failure using partial pressure of oxygen (PaO₂) and fraction of inspired oxygen (FiO₂) is defined by a partial pressure of oxygen/fraction of inspired oxygen ratio (PaO₂/FiO₂) ≤ 300 mmHg or a respiratory rate (RR) ≥ 25/min
* Informed consent obtained

Exclusion Criteria:

* Hemodynamic instability requiring vasopressors
* Altered mental status Glasgow Coma Scale (GCS < 13)
* Contraindication to NIV or HVNI (facial trauma, recent upper airway surgery)
* Do-Not-Intubate (DNI) order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Failure Within 48 Hours | 48 hours after randomization
  Treatment failure is defined as the occurrence of either endotracheal intubation or death within 48 hours following randomization. This composite endpoint assesses the immediate efficacy of the assigned respiratory support modality-High-Velocity Nasal Insufflation (HVNI) or Noninvasive Ventilation (NIV)-in preventing rapid clinical deterioration in patients with acute exacerbations of community-acquired pneumonia (CAP) accompanied by hypoxemic respiratory failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M. Shaddad, MD, Principal Investigator — Assiut University; Aliae A. Hussien, MD, Principal Investigator — Assiut University
Locations (1):
- Assuit University, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Plan Description: De-identified individual participant data supporting the primary and secondary outcomes, along with accompanying data dictionaries and the statistical analysis plan, will be made available in accordance with Assiut University's institutional data-sharing policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be accessible 6-36 months after publication
Access Criteria: Data will be accessible 6-36 months after publication to qualified researchers upon submission of a study proposal, approval by the University Research Ethics Committee, and execution of a data-use agreement.